CLINICAL TRIAL: NCT01341821
Title: Influences of Leadership Style on Team Climate for Quality
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Liang-Ming Lee, Superintendent Office, Wanfang Hospital
Other Study IDs: 99023
Record Dates: First submitted 2011-04-24; First posted 2011-04-26 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Leadership Style
Keywords: Leadership Style; Team Climate

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to discuss how different personalities of leaders and employees result in the effect of quality and efficiency in different organizational climate and also how the leadership style of different leaders affect the organizational climate. The investigators hope that this study will improve the key factor of quality and efficiency among leaders. Besides, the investigators want to provide the reference of quality control for the groups of healthcare quality in order to avoid unnecessary time and costs and achieve the goal of improvement quality.

DETAILED DESCRIPTION:
The specific purpose of this study is the following:

1. to discuss the relationship of organizational climate due to different leadership styles.
2. to discuss the relationship of quality efficiency due to different organizational climates.
3. to discuss the relationship of quality efficiency due to different leadership styles.

ELIGIBILITY:
Inclusion Criteria:

* employees in the hospitals

Exclusion Criteria:

* none employees in the hospitals

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: employees in the hospitals
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-05; Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Ming Lee, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan